CLINICAL TRIAL: NCT07275957
Title: Study of the Effects of Implementing Dietary-nutritional Strategies and an Exercise Program at the Physical, Physiological, and Psychological Level in Women With a History of Breast Cancer.
Brief Title: Combined Nutrition and Exercise Interventions in Women With Breast Cancer History
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alicante (Other)
Responsible Party: Principal Investigator, Prof. Dr. Alejandro Martínez-Rodríguez, Full Professor of Health Sciences, University of Alicante
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UA-2025-06-13
Record Dates: First submitted 2025-11-25; First posted 2025-12-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer Survivors
Keywords: Breast cancer survivors; Exercise intervention; Nutritional intervention; Mediterranean diet; Physical rehabilitation; Quality of life; Body composition; Strength training; Aerobic exercise; Combined training; Lifestyle modification

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of six parallel intervention arms (control, Mediterranean diet, strength training, endurance training, combined training, or Mediterranean diet plus combined training). The interventions will be carried out simultaneously over 12 weeks, with pre- and post-intervention assessments to evaluate changes in physical, physiological, and psychological parameters.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 - Control Group (No Intervention): Participants will not receive any specific dietary or exercise intervention. They will be asked to maintain their usual lifestyle and dietary habits during the 12-week study period. General health recommendations based on national guidelines will be provided at baseline.
- Arm 2 - Mediterranean Diet Group (MD) (Experimental): Participants will receive individualized nutritional counseling promoting adherence to a Mediterranean dietary pattern, emphasizing fruits, vegetables, legumes, whole grains, olive oil, nuts, fish, and moderate dairy intake. Processed and high-sugar foods will be limited. Dietitians will provide personalized follow-up and adjustments every two weeks to ensure adherence.
  Interventions: Behavioral: Mediterranean Diet Counseling
- Arm 3 - Strength Training Group (ST) (Experimental): Participants will perform a 12-week supervised resistance training program focused on improving muscular strength and functional capacity. Sessions will be conducted three times per week, lasting approximately 60 minutes, and include major muscle groups using elastic bands, free weights, and bodyweight exercises. Training load will progressively increase according to individual capacity.
  Interventions: Behavioral: Supervised Strength Training Program
- Arm 4 - Endurance Training Group (ET) (Experimental): Participants will follow a structured aerobic exercise program consisting of walking, cycling, or treadmill sessions three times per week for 12 weeks. The intensity will be moderate (60-75% of estimated maximal heart rate), gradually progressing as tolerated. The goal is to enhance cardiorespiratory fitness and overall endurance.
  Interventions: Behavioral: Supervised Endurance Training Program
- Arm 5 - Combined Training Group (CT) (Experimental): Participants will perform both strength and aerobic training during the 12-week intervention. Each session (3 per week, 60-70 minutes) will include resistance exercises targeting major muscle groups followed by aerobic activity at moderate intensity. The program aims to improve both muscular and cardiovascular performance synergistically.
  Interventions: Behavioral: Combined Strength and Endurance Training Program
- Arm 6 - Mediterranean Diet plus Combined Training Group (MD+CT) (Experimental): Participants will simultaneously receive the Mediterranean Diet counseling and participate in the Combined Training program for 12 weeks. The objective is to assess the synergistic effects of diet and exercise on physical, physiological, and psychological health in breast cancer survivors.
  Interventions: Behavioral: Combined Mediterranean Diet and Exercise Program

INTERVENTIONS:
Behavioral: Mediterranean Diet Counseling — Individualized nutritional counseling based on Mediterranean diet principles, emphasizing the intake of fruits, vegetables, legumes, whole grains, nuts, olive oil, and fish, while reducing red meat, processed foods, and added sugars. Sessions will be held biweekly to ensure adherence and promote long-term dietary behavior change.
  Arms: Arm 2 - Mediterranean Diet Group (MD)
Behavioral: Supervised Strength Training Program — A structured resistance exercise program performed three times per week for 12 weeks. Each 60-minute session will include exercises for major muscle groups using elastic bands, dumbbells, or body weight, progressively increasing intensity to improve muscle strength and endurance.
  Arms: Arm 3 - Strength Training Group (ST)
Behavioral: Supervised Endurance Training Program — A structured aerobic exercise program consisting of walking, cycling, or treadmill training three times per week for 12 weeks. Exercise intensity will range from 60% to 75% of the estimated maximal heart rate, progressively adjusted to enhance cardiovascular fitness and fatigue resistance.
  Arms: Arm 4 - Endurance Training Group (ET)
Behavioral: Combined Strength and Endurance Training Program — A combined exercise protocol including both resistance and aerobic components within each 60-70-minute session, three times per week for 12 weeks. Strength exercises will precede moderate-intensity aerobic work to improve overall physical performance and functional capacity.
  Arms: Arm 5 - Combined Training Group (CT)
Behavioral: Combined Mediterranean Diet and Exercise Program — Comprehensive lifestyle intervention combining Mediterranean diet counseling with the supervised combined training program. Participants will receive individualized diet plans and attend three supervised exercise sessions per week. The intervention targets improvements in body composition, physical fitness, and emotional well-being.
  Arms: Arm 6 - Mediterranean Diet plus Combined Training Group (MD+CT)

SUMMARY:
This study aims to evaluate the effects of a combined dietary-nutritional and physical exercise intervention on physical, physiological, and psychological outcomes in women who are breast cancer survivors. Participants will be randomly assigned to different intervention groups involving dietary modification, exercise training, or their combination, compared to a control group. The program will last 12 weeks and will include pre- and post-intervention assessments of body composition, metabolic parameters, functional capacity, and quality of life.

The primary goal is to assess improvements in physical fitness, body composition, and emotional well-being, as well as to identify potential synergistic effects of combined interventions in this population.

DETAILED DESCRIPTION:
Breast cancer survivors often experience long-term physical and psychological side effects derived from treatment, such as fatigue, loss of muscle mass, metabolic alterations, and reduced quality of life. Lifestyle interventions involving nutrition and exercise have demonstrated significant potential to mitigate these effects and promote overall recovery.

This randomized controlled clinical trial will include adult female breast cancer survivors who have completed their primary oncological treatment. Participants will be divided into six parallel groups:

1. Control group - no intervention.
2. Mediterranean diet group (MD) - individualized nutritional plan based on Mediterranean dietary patterns.
3. Strength training group (ST) - supervised resistance exercise sessions.
4. Endurance training group (ET) - supervised aerobic exercise sessions.
5. Combined training group (CT) - combination of strength and endurance training.
6. Combined diet and exercise group (MD+CT) - simultaneous application of Mediterranean diet and combined training.

The intervention will last 12 weeks, during which participants in the intervention groups will attend supervised sessions and receive continuous nutritional guidance. Assessments will be performed at baseline and after 12 weeks, including anthropometric and body composition analysis, metabolic and inflammatory markers, physical fitness testing, dietary intake, and psychological well-being scales.

This study seeks to identify the most effective strategy-dietary, physical, or combined-for improving health outcomes, functionality, and emotional recovery in breast cancer survivors, contributing to the development of comprehensive post-treatment rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 30 to 65 years.
* Previous diagnosis of breast cancer (stages I-III) confirmed by medical records.
* Completion of primary oncological treatment (surgery, radiotherapy, chemotherapy, and/or hormone therapy) at least 3 months before enrollment.
* Absence of active cancer or evidence of recurrence.
* Medical clearance to perform physical exercise.
* Willingness to participate in dietary and/or exercise interventions for 12 weeks.
* Ability to attend evaluation and intervention sessions and comply with study procedures.
* Signed written informed consent.

Exclusion Criteria:

* Active cancer, metastasis, or ongoing chemotherapy or radiotherapy.
* Severe cardiovascular, respiratory, renal, hepatic, or metabolic disease that contraindicates exercise.
* Musculoskeletal or neurological conditions limiting participation in physical activity.
* Severe psychiatric disorders or cognitive impairment affecting adherence to the intervention.
* Current participation in another clinical trial or structured lifestyle intervention.
* Use of dietary supplements, appetite regulators, or pharmacological agents affecting metabolism during the study period.
* Pregnancy, breastfeeding, or intention to become pregnant during the study.
* Inability to comply with the intervention schedule or follow-up assessments.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fat-Free Mass (kg) | Baseline and Week 12
  To evaluate changes in fat-free mass after the 12-week intervention, measured by bioimpedance analysis (BIODY XPERT ZM).

SECONDARY OUTCOMES:
Change in Fat Mass (%) | Baseline and Week 12
  To assess changes in total body fat percentage using bioimpedance analysis.
Change in Body Weight (kg) | Baseline and Week 12
  To determine body weight variation during the 12-week intervention.
Change in Body Mass Index (kg/m²) | Baseline and Week 12
  To evaluate changes in BMI calculated as weight divided by height squared.
Change in Waist Circumference (cm) | Baseline and Week 12
  To assess central adiposity changes by measuring waist circumference.
Change in Handgrip Strength (kg) | Baseline and Week 12
  To evaluate upper-body muscular strength using a digital hand dynamometer.
Change in Lower-Limb Strength (kg) | Baseline and Week 12
  To assess lower-limb strength through isometric tests using a load cell or force platform.
Change in Functional Capacity (6-Minute Walk Test Distance, m) | Baseline and Week 12
  To evaluate cardiorespiratory endurance using the 6-minute walk test.
Change in Balance Performance | Baseline and Week 12
  To assess dynamic balance and postural control
Change in Flexibility (Sit-and-Reach Test, cm) | Baseline and Week 12
  To evaluate flexibility of the posterior chain through the sit-and-reach test.
Change in Maximal Oxygen Uptake (VO₂max, mL/kg/min) | Baseline and Week 12
  To determine changes in aerobic capacity using an incremental treadmill test with indirect calorimetry (METALYZ-ERR 3 B-R3 spirometer).
Change in Total Cholesterol (mg/dL) | Baseline and Week 12
  To evaluate lipid profile variations by measuring total cholesterol concentration.
Change in HDL Cholesterol (mg/dL) | Baseline and Week 12
  To assess cardioprotective lipid changes.
Change in LDL Cholesterol (mg/dL) | Baseline and Week 12
  To measure changes in LDL cholesterol levels.
Change in Triglycerides (mg/dL) | Baseline and Week 12
  To determine variations in triglyceride concentration.
Change in Fasting Glucose (mg/dL) | Baseline and Week 12
  To assess metabolic health by measuring fasting plasma glucose.
Change in C-Reactive Protein (mg/L) | Baseline and Week 12
  To evaluate systemic inflammation using CRP levels.
Change in Interleukin-6 (pg/mL) | Baseline and Week 12
  To measure inflammatory status via IL-6 concentration.
Change in Fatigue (FACIT-F Questionnaire Score) | Baseline and Week 12
  Description: Fatigue will be assessed using the Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F). This questionnaire consists of 13 items rated on a 5-point Likert scale ranging from 0 ("not at all") to 4 ("very much"), reflecting fatigue experienced during the past 7 days. The total score is calculated by summing the item scores (after reverse scoring where applicable). Range: 0-52. Interpretation: Higher scores indicate less fatigue and therefore a better functional status, while lower scores reflect greater fatigue severity.
Change in Sleep Quality (PSQI Total Score) | Baseline and Week 12
  Description: Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a 19-item self-reported questionnaire that evaluates sleep quality and disturbances over the previous month. The items are grouped into seven components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction), each scored from 0 to 3. The global PSQI score is the sum of the components (range 0-21). Range: 0-21. Interpretation: Higher scores indicate poorer sleep quality.
Change in Physical Activity Level (IPAQ Total Score) | Baseline and Week 12
  Description: Physical activity levels will be evaluated using the International Physical Activity Questionnaire - Short Form (IPAQ-SF), which records the frequency and duration of walking, moderate, and vigorous activities over the past 7 days. The results are expressed as total metabolic equivalent minutes per week (MET-min/week) and can be categorized into three levels: low, moderate, or high activity. Range: 0 to unlimited MET-min/week. Interpretation: Higher scores indicate higher physical activity levels.
Change in Dietary Adherence (Mediterranean Diet Adherence Screener Score) | Baseline and Week 12
  Description: Adherence to the Mediterranean diet will be assessed using the PREDIMED Questionnaire, a validated 14-item questionnaire evaluating key dietary habits such as olive oil use, fruit and vegetable consumption, fish intake, and limitation of red meat and sweets. Each affirmative answer scores 1 point, yielding a total score from 0 (minimal adherence) to 14 (maximal adherence). Range: 0-14. Interpretation: Higher scores indicate better adherence to the Mediterranean dietary pattern.

CONTACTS AND LOCATIONS:
Locations (1):
- European Institute Of Exercise and Health, Elche, Alicante, Spain